CLINICAL TRIAL: NCT00776581
Title: A Ten-year Practice of Labor Pain Control in China
Brief Title: Ten-year Practice of Labor Pain Control in China
Acronym: POPIC
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Other Study IDs: NMU-FY2008-MZ013; NJFY081005
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Labor Pain
Keywords: Combined spinal-epidural analgesia; Patient-controlled analgesia; Epidural analgesia
MeSH Terms: conditions — Labor Pain | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Records regarding combined spinal-epidural analgesia (CSEA) with patient-controlled analgesia (PCA) pump
  Interventions: Procedure: CSEA with PCA
- 2: Records regarding combined spinal-epidural analgesia with intermittent bolus injection (IBI)
  Interventions: Procedure: CSEA with IBI
- 3: Records regarding epidural analgesia (EA) with patient-controlled pump
  Interventions: Procedure: EA with PCA
- 4: Records regarding epidural analgesia with intermittent bolus injection
  Interventions: Procedure: EA with IBI

INTERVENTIONS:
Procedure: CSEA with PCA — Records regarding combined spinal-epidural analgesia with patient-controlled pump
  Groups: 1
Procedure: CSEA with IBI — Records regarding combined spinal-epidural analgesia with intermittent bolus injection
  Groups: 2
Procedure: EA with PCA — Records regarding epidural analgesia with patient-controlled pump
  Groups: 3
Procedure: EA with IBI — Records regarding epidural analgesia with intermittent bolus injection
  Groups: 4

SUMMARY:
Since 1999, labor pain control has being performed in China, and the initial time of analgesia is at the cervix >= 2 cm. Meanwhile, American Society of Obstetrics & Gynecology recommended that the labor analgesia with neuraxial block should be performed at the cervix >= 4 cm in 2002. After that, the threshold has been revised to at least >= 2 cm in 2006 by the Society. However, in China, the practice of labor analgesia with neuraxial block has being performed for over seven years. Up until now, the practice has being experienced during this ten-year period at the cervix around 1 cm. The investigators hypothesized that labor pain control in different stages had different characteristics and had different influence on patients short- and long-lasting outcomes. This study is mainly investigating different labor analgesia procedures in different stages since the initiation of the practice in 1999, and assessing their influence on the outcomes to display the trajectory of development of labor analgesia in China of which might fit to the the whole process of the study of labor analgesia throughout the world. All these were done by analyzing the data records since from January 1999 to December 2008.

ELIGIBILITY:
Inclusion Criteria:

* Parturients used labor analgesia

Exclusion Criteria:

* Following criteria were based on the records of information received from the ten-year practice screened by investigators:

  1. Chronic pain and psychiatric diseases records
  2. Participants younger than 18 years or older than 45 years
  3. Alcohol addictive or narcotic dependent patients were excluded for their influence on the analgesic efficacy of the epidural analgesics
  4. Subjects with a nonvertex presentation or scheduled induction of labor
  5. Diagnosed diabetes mellitus and pregnancy-induced hypertension
  6. Twin gestation and breech presentation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All parturients delivered in the investigator's institution since from January 1999 to December 2008
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Rate of cesarean delivery | Analgesia initiation to successful vaginal delivery

SECONDARY OUTCOMES:
Rate of instrument-assisted delivery | Analgesia initiation to successful vaginal delivery
Indications of cesarean delivery | Analgesia initiation to cesarean section
Maternal Visual Analog Scale (VAS) rating of pain | Prior to analgesia, latent phrase, active phrase, second stage of labor, posterior to vaginal delivery
Duration of analgesia | Initiation of analgesia to the disappearance of sensory block
Maternal satisfaction with analgesia | At the end of the vaginal delivery
Maternal oral temperature | Analgesia initiation to successful vaginal delivery
Use of oxytocin after analgesia | After analgesia to vaginal delivery
Low back pain at 3 months after vaginal delivery | At the third month after vaginal delivery
Breastfeeding success at 6 weeks after vaginal delivery | At the sixth week after successful delivery
Neonatal one-minute Apgar scale | At the first minute of baby was born
Neonatal five-minute Apgar scale | At the fifth minute of baby was born
Incidence of maternal side effects | Analgesia initiation to successful vaginal delivery
Umbilical-cord gases analysis | At the time baby was born

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China